CLINICAL TRIAL: NCT03732482
Title: A Phase II/III Study of Non Small Cell Lung Cancer Patient With/Without Synchronous Oral Temozolomide Capsules Combine With Intensity Modulated Radiation Therapy With Simultaneous Integrated Boost With Hippocampus Protection
Brief Title: Temozolomide Combine With Intensity Modulated Radiation Therapy With Simultaneous Integrated Boost for Non Small Cell Lung Cancer Brain Metastases
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Haihua Yang, head of department of Radiation Oncology,chief physician,, Taizhou Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YHH-201807
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Non Small Cell Lung Cancer Metastatic
MeSH Terms: interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT groups (Placebo Comparator): participants was given radiotherapy only,50Gy in 10 fractions over 2 weeks to metastases synchronously with 25Gy WBRT
  Interventions: Device: radiotherapy
- Drug plus RT groups (Experimental): Temozolomide capsules(Jiangsu tasly diyi pharmaceutical Co.,Ltd) Oral Temozolomide capsules 75mg/m2 begins on day 1 and continues until completion of radiotherapy.
  Interventions: Drug: Temozolomide capsules

INTERVENTIONS:
Drug: Temozolomide capsules — Temozolomide capsules(Jiangsu tasly diyi pharmaceutical Co.,Ltd) Oral Temozolomide capsules 75mg/m2 begins on day 1 and continues until completion of radiotherapy.
  Arms: Drug plus RT groups
Device: radiotherapy — Intensity Modulated Radiation Therapy With Simultaneous Integrated Boost
  Arms: RT groups

SUMMARY:
With the improvement of systemic therapeutic effect(especially in the population with driver gene mutation), the incidence of brain metastases had significantly increased. Conventional Whole Brain radiotherapy(WBRT) was less effective, the stereotactic radiosurgery(SRS) technique had improve the local efficacy for 1-3 lesions, but the probability of intracranial recurrence was increased, Intensity Modulated Radiation Therapy With Simultaneous Integrated Boost(SIB-IMRT) is a new radiotherapy technology, Giving a standard radiation dose of whole brain ,at the same time can boost the high-risk region in target, So that it can significantly shorten the treatment time, at the same time can improve the local control rate of brain metastases. In the aspect of normal tissue protecting, SIB was better than WBRT plus SRS sequential treatment pattern. 30Gy to the whole brain had a negative effects on cognitive function, the investigators previous study found that 25Gy to the whole brain while the tumor bed Simultaneous push to 50Gy was safe and effective, while reducing the impact on cognitive function. Hippocampus is a part of the brain located in the temporal lobe, Mainly responsible for long-term memory storage conversion and orientation. Many investigators point out that hippocampus is the main commander of neurocognitive function, Reduce the dose of hippocampus can significant improve the neurocognitive function. Temozolomide capsule is an anti-tumor alkylation agent for glioblastoma multiforme and anaplastic astrocytoma. In recent years, some researchers find that Temozolomide capsules combine with radiotherapy such as SRS, WBRT or The two combined, can improve Objective response(OR) and prolong the Progress Free Survival(PFS),while with tolerable therapeutic toxicity. In order to better reduce the impact on cognitive function and improve the local control rate, the investigators present this trial, under the SIB-IMRT technique, the investigators want to explore the effect of temozolomide in brain metastasis of non-small cell lung cancer with the hippocampal protection technology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have an estimated survival of at least 4 weeks
2. Karnofsky Performance Status Scale (KPS) of 60-100.
3. Patients' laboratory values had to meet these restrictions: hemoglobin>8 g/dL, platelets>70*109/L, white blood cells>4*109/L.
4. Patients must sign a study specific informed consent form prior to study entry

Exclusion Criteria:

1. Patients had major medical illnesses or psychiatric impairments which will prevent completion of the protocol therapy
2. had received previous brain irradiation
3. could not be regularly followed
4. with leptomeningeal involvement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
OS | Duration of time from the start of therapy 3 years or until time of death, whichever occurs first
  overall survival

SECONDARY OUTCOMES:
iPFS | Duration of time from the start of therapy to the time of intracranial disease progression, assessed up to 3 years
  intracranial Progress Free Survival
MMSE scores | up to 2 years
  mini mental state examination,The MMSE scores included 11 questions and was consisted of orientation to time (5 scores), orientation to place (5 scores), registration (3 scores), attention and calculation (5 scores), recall (3 scores), langue (2 scores), repetition (1 scores), complex commands (6 scores). The minimum score was 0, The maximum score was 30.
overall response rate | Up to 1 month
  use RECIST 1.1 version

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhu, MD, Principal Investigator — Taizhou Hospital, Wenzhou Medical University